CLINICAL TRIAL: NCT04387370
Title: Comparison of Single and Double Hem-o-log Clips in Laparoscopic Appendectomy
Brief Title: The Use of the Hem-o-lok Clip in Appendectomy: Single or Double?
Status: Completed | Type: Observational
Sponsor: Ulas Aday (Other Government)
Responsible Party: Sponsor-Investigator, Ulas Aday, Assistant professor, Kartal Kosuyolu Yuksek Ihtisas Education and Research Hospital
Organization: Kartal Kosuyolu Yuksek Ihtisas Education and Research Hospital (Other Government)
Other Study IDs: 'KartalH'
Record Dates: First submitted 2020-04-29; First posted 2020-05-13 (Actual); Last update posted 2023-04-19 (Actual); Status verified 2023-04

CONDITIONS: Acute Appendicitis
Keywords: Laparoscopic appendectomy; Hem-o-lok clip; stump closure
MeSH Terms: conditions — Appendicitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Stump safety is provided by different methods in laparoscopic appendectomy. Stapler use, binding with endoloop and nonabsorbable clip are the most common methods. Although the stapler is safe, it creates a significant cost increase. In connecting with the endoloop, the learning curve and surgical time are longer. Nonabsorbable clip application which has been used recently; Urethra was also used in appendectomy after its safety has been proven by large studies to close cystic ducts and vascular structures. Its advantages such as low cost, no need for a learning curve and shortening the surgical time have increased the frequency of use.In this prospective observational study; It will be aimed to investigate the effects of stump closure methods applied in laparoscopic appendectomy on short-term clinical results. In addition, the factors that determine the surgeon's stump closure method and cost results will be tried to be determined.

DETAILED DESCRIPTION:
Detailed explanation will be made later if necessary.

ELIGIBILITY:
Inclusion Criteria

* diagnosis of acute appendicitis
* Performing laparoscopic surgery
* Patients with an ASA score of I-II-III

Exclusion Criteria:

* Appendectomies with the patient's refusal to participate in the study
* Open surgery
* Primary pathology without appendicitis

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Patients over 18 years old
Study Population: Patients operated on for acute appendicitis
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-04-18 (Actual)

PRIMARY OUTCOMES:
Is it safe to close the appendix stump with a single hem-o-lok clip? | one year
  Complications of patients using single and double clips will be compared according to Clavien-Dindo scoring system.

SECONDARY OUTCOMES:
The effect of single and double hem-o-lok clips on cost in laparoscopic appendectomy | one week
  With the use of a single clip, surgery costs are expected to be less in dollars.Student's t-test will be used for cost analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Abdullah Oğuz, MD, Principal Investigator — Dicle University Medical of School; Ulaş Aday, MD, Study Chair — Dicle University Medical of School; Mehmet veysi Bahadır, MD, Study Director — Dicle University Medical of School
Locations (1):
- Dicle University Medical of School, Department of Gastrointestinal Surgery, Diyarbakır, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Since there are no plans yet, planning will be done later.

REFERENCES:
- [Derived] Aday U, Cetin E, Kafadar MT, Oguz A, Bahadir MV, Ulger BV, Gedik E, Girgin S, Yilmaz M. Single versus double Hem-o-lok clips to secure the apendiceal stump during laparoscopic appendectomy: a prospective randomized multicentric clinical trial. Langenbecks Arch Surg. 2024 Mar 8;409(1):89. doi: 10.1007/s00423-024-03281-4. PMID 38457041